CLINICAL TRIAL: NCT00481975
Title: A Randomized, Double-Bind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multicenter Study to Assess Efficacy and Safety of Rimonabant 20 mg Versus Placebo on Weight Loss and Frequency of Binge Episodes in Obese Patients With Food Craving
Brief Title: Efficacy and Safety of Rimonabant on Weight Loss and Frequency of Binge Episodes in Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT3801
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Obesity; Eating Disorders
Keywords: binge eating; eating disorders; obesity
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders; Bulimia | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary objective is to assess the effect of rimonabant compared to placebo on weight loss over a period of 6 months when prescribed with a mild hypocaloric diet in obese patients with binge eating disorder.

The secondary objectives are:

* to assess the effect of rimonabant on the number of binge episodes per week, to assess the effect of rimonabant on eating behavior using the Binge Eating Scale (BES) and Three Factor Eating Questionnaire (TFEQ),
* to evaluate the safety and tolerability of rimonabant over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥30 to ≤45 kg/m²
* Diagnosis of eating disorder using The Questionnaire on Eating and Weight Patterns (QEWP-R) for diagnosing Eating Behaviors

Exclusion Criteria:

* History of surgical procedures for weight loss
* Treatment with anti-obesity drugs within 3 months prior to screening visit
* Presence or history of Diagnostic and Statistical Manual of Mental Disorders (4th edition)(DSM IV) bulimia or anorexia nervosa

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline to Day 180 visit

SECONDARY OUTCOMES:
Efficacy: binge eating episodes, BES score, TFEQ dimensions, waist circumference, Body Mass Index
Safety: clinical examination, vital signs, adverse events, Hospital Anxiety and Depression (HAD) scale

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Derived] Pataky Z, Gasteyger C, Ziegler O, Rissanen A, Hanotin C, Golay A. Efficacy of rimonabant in obese patients with binge eating disorder. Exp Clin Endocrinol Diabetes. 2013 Jan;121(1):20-6. doi: 10.1055/s-0032-1329957. Epub 2012 Nov 12. PMID 23147209